CLINICAL TRIAL: NCT04863144
Title: Effect of CYP3A4 and CYP2C8 Activity on Pharmacokinetics of Paclitaxel, Correlation With Adverse Events in Cancer Patients With and Without Liver Impairment
Brief Title: Pharmacokinetics of Paclitaxel in Correlation With Adverse Events in Cancer Patients With and Without Liver Impairment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU MD 8/2020
Record Dates: First submitted 2021-04-21; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Liver Diseases
Keywords: Paclitaxel; Pharmacokinetics; Egypt
MeSH Terms: conditions — Liver Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood samples — Plasma concentrations of paclitaxel and its metabolites will be obtained during the first treatment cycle. The samples for paclitaxel analysis will be collected in ethylenediamine tetraacetic acid tubes at 7-time points: just before infusion, in the middle of the infusion, at the end of infusion, at 1, 2, 4 and 6 hours post-infusion.

SUMMARY:
The study aims to assess the pharmacokinetics of paclitaxel and its two major metabolites in patients with normal and impaired liver functions.

DETAILED DESCRIPTION:
population pharmacokinetic study in patients with normal or impaired liver functions, receiving paclitaxel for cancer treatment.

40 Patients with histologically confirmed solid tumors will be enrolled in the study:

* 20 patients have normal liver functions as defined by transaminase < 2.6 x ULN and bilirubin values < 1.26 x ULN.
* 20 patients with liver impairment as defined by transaminase 2.6 - 10 x ULN and bilirubin values 1.26 - 5 x ULN.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven non haematopoietic malignancy (ovarian, breast and lung cancer).
* Age between 18 and 70 years
* At least a 4-week interval between the last dose of previous chemotherapy protocol and registration (6 weeks in case of treatment with carboplatin).
* Glomerular filtration rate > 60 ml/min
* An Eastern Cooperative Oncology Group performance status 0-2, a life expectancy of > 12 weeks, adequate bone marrow function [absolute neutrophil count (ANC) ≥ 1 X 109 and platelets ≥ 100 X 109]
* Patient accessible for treatment and follow-up and written informed consent.

Exclusion Criteria:

* Prior treatment with paclitaxel or other taxanes.
* Pre-existing motor or sensory neurotoxicity > grade 2 according to World Health Organization (WHO) criteria.
* Active infection or other serious underlying medical condition (including prior allergic reactions to Paclitaxel or the drug's constituents), dementia or significantly altered mental status, symptomatic brain or liver metastases, history of atrial or ventricular arrhythmias or congestive heart failure even if medically controlled, history of clinical and electrocardiographically documented myocardial infarction.
* Simultaneous use of any medication, dietary supplements, or other compounds known to inhibit affect the pharmacokinetics of paclitaxel.
* Patients with difficult blood sampling.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 Patients with histologically confirmed solid tumors and are going to receive paclitaxel
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
plasma concentrations of paclitaxel | predose till 6 hours post infusion of paclitaxel
  determination of plasma concentration and pharmacokinetic analysis of paclitaxel
plasma concentrations of 6-α-hydroxypaclitaxel | predose till 6 hours post infusion of paclitaxel
  determination of plasma concentration and pharmacokinetic analysis of 6-α-hydroxypaclitaxel
plasma concentrations of 3'-p-hydroxypaclitaxel | predose till 6 hours post infusion of paclitaxel
  determination of plasma concentration and pharmacokinetic analysis of 3'-p-hydroxypaclitaxel

SECONDARY OUTCOMES:
Probing CYP 3A4 activity | predose till 6 hours post infusion of paclitaxel
  metabolite ratio of 6-α-hydroxypaclitaxel/paclitaxel
Probing CYP 2C8 activity | predose till 6 hours post infusion of paclitaxel
  metabolite ratio of 3'-p-hydroxypaclitaxel/paclitaxel
Incidence of adverse effects | baseline ( before first dose) till 100 days after the first dose
  Complete blood count, liver functions and neuropathy evaluation (according to Common Terminology Criteria for Adverse Events (CTCAE), version 5) will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Nour-Eldin, Professor, Study Director — Pharmacology Department - Faculty of Medicine - Ain Shams University; Khaled Abdel-Aziz, MD, Study Director — Oncology Department - Faculty of Medicine - Ain Shams University
Locations (1):
- El Demerdash Oncology Hospital, Cairo, Abbasia, Egypt